CLINICAL TRIAL: NCT06048094
Title: 18F-Fluciclovine PET Amino Acid Evaluation of Brain Metastasis Treated With Stereotactic Radiosurgery (FACILITATE)
Brief Title: 18F-Fluciclovine PET Amino Acid Evaluation of Brain Metastasis Treated With Stereotactic Radiosurgery
Acronym: FACILITATE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baptist Health South Florida (Other)
Collaborators: Blue Earth Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-KOT-003
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Brain Metastases; Brain Metastases, Adult; Brain Cancer
Keywords: stereotactic radiosurgery; 18F-flucicloivine; PET imaging
MeSH Terms: conditions — Brain Neoplasms | interventions — fluciclovine F-18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 18F-Fluciclovine PET Imaging (Experimental): Participants will undergo a 18F-fluciclovine PET scan at the time of their SRS planning magnetic resonance imaging (MRI). Then participants will undergo single-fraction SRS as standard of care (SOC). A second 18F-fluciclovine PET scan will be completed 8 weeks (± 2 weeks) after SRS.
  Interventions: Drug: 18F fluciclovine

INTERVENTIONS:
Drug: 18F fluciclovine — Participants will receive 5-mCi dose (± 20%) of 18F-fluciclovine intravenously as a bolus injection immediately prior to PET data acquisition. PET data will be collected in list mode up to 25 minutes post-injection. PET images will be reconstructed in two ways: as a standard static image of data acquired between 10 to 20 minutes post-injection, and as a dynamic series of four 5-minute frames between 5 to 25 minutes post-injection to allow for motion assessment and correction and time-dependent observations.
  Other Names: Axumin; 18F-FACBC; (1r, 3r)-1-amino-3[18F] fluorocyclobutane-1-carboxylic acid

SUMMARY:
This is a pilot imaging study in participants treated with stereotactic radiosurgery (SRS) to treat brain metastasis. The purpose of this study is to see whether 18F-Fluciclovine positron emission tomography (PET) can be used as a biomarker to measure response or progression of brain metastasis after SRS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer with radiographic finding of brain metastasis
* Any number of brain metastasis, with all lesions ≤ 2 cm in maximum dimension
* Planned treatment with SRS as per the treating physician team
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Individuals of reproductive potential need to employ two highly effective and acceptable forms of contraception for at least 4 weeks prior to screening and agree to use such a method during study participation up to an additional 1 week following the last 18F-fluciclovine PET

Exclusion Criteria:

* Prior anaphylactic reaction to 18F-fluciclovine
* Radiographic evidence of leptomeningeal disease
* Prior whole-brain radiation therapy
* Inability to undergo MRI (e.g., due to safety reasons, such as presence of a pacemaker)
* Pregnant or positive serum pregnancy test within 14 days of registration
* Individuals expecting to be breastfeeding at the time of 18F-fluciclovine and unwilling to stop breast-feeding for 24 hours. Temporary cessation of breastfeeding for 24 hours after the time of imaging is allowed.
* Major medical illness or psychiatric/cognitive impairments, which in the investigator's opinion, will prevent completion of protocol and/or preclude informed consent*

  * A legally authorized representative (LAR) may consent on a potential participant's behalf in the case of cognitive impairment, if in the investigator's opinion, that impairment would not prevent completion of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change in Standardized Uptake Value (SUV)-peak | 8 weeks
  Each 18F-fluciclovine PET will undergo quantitative image analysis by the study nuclear medicine physician. The lesion on each PET will be correlated with the lesion on the corresponding contrast-enhanced MRI and will be delineated. The SUVpeak will be calculated for the pre-SRS and post-SRS imaging studies, as well as the percent change from pre to post will be calculated. Assuming SRS reduces the tumor size, a negative percent change (decrease) is expected.
Change in SUVmean | 8 weeks
  Each 18F-fluciclovine PET will undergo quantitative image analysis by the study nuclear medicine physician. The lesion on each PET will be correlated with the lesion on the corresponding contrast-enhanced MRI and will be delineated. The SUVmean will be calculated for the pre-SRS and post-SRS imaging studies, as well as the percent change from pre to post will be calculated. Assuming SRS reduces the tumor size, a negative percent change (decrease) is expected.
Change in SUVmax | 8 weeks
  Each 18F-fluciclovine PET will undergo quantitative image analysis by the study nuclear medicine physician. The lesion on each PET will be correlated with the lesion on the corresponding contrast-enhanced MRI and will be delineated. The SUVmax will be calculated for the pre-SRS and post-SRS imaging studies, as well as the change from pre to post will be calculated. Assuming SRS reduces the tumor size, a negative percent change (decrease) is expected.

SECONDARY OUTCOMES:
Tumor Control | 12 months
  Each lesion will be followed from pre-treatment PET to local failure or retreatment; death; lost-to follow-up, discontinuation, or withdrawal; or end of study. Local failure is defined as disease progression according to Response Assessment in Neuro-Oncology (RANO) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Rupesh Kotecha, M.D., Principal Investigator — Miami Cancer Institute at Baptist Health, Inc.
Locations (1):
- Miami Cancer Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galldiks N, Langen KJ. Amino acid PET in neuro-oncology: applications in the clinic. Expert Rev Anticancer Ther. 2017 May;17(5):395-397. doi: 10.1080/14737140.2017.1302799. Epub 2017 Mar 11. No abstract available. PMID 28277832
- [Background] Doi Y, Kanagawa M, Maya Y, Tanaka A, Oka S, Nakata N, Toyama M, Matsumoto H, Shirakami Y. Evaluation of trans-1-amino-3-18F-fluorocyclobutanecarboxylic acid accumulation in low-grade glioma in chemically induced rat models: PET and autoradiography compared with morphological images and histopathological findings. Nucl Med Biol. 2015 Aug;42(8):664-72. doi: 10.1016/j.nucmedbio.2015.04.008. Epub 2015 May 7. PMID 26022202
- [Background] Parent EE, Patel D, Nye JA, Li Z, Olson JJ, Schuster DM, Goodman MM. [18F]-Fluciclovine PET discrimination of recurrent intracranial metastatic disease from radiation necrosis. EJNMMI Res. 2020 Dec 7;10(1):148. doi: 10.1186/s13550-020-00739-6. PMID 33284388
- [Background] Wakabayashi T, Hirose Y, Miyake K, Arakawa Y, Kagawa N, Nariai T, Narita Y, Nishikawa R, Tsuyuguchi N, Fukami T, Sasaki H, Sasayama T, Kondo A, Iuchi T, Matsuda H, Kubota K, Minamimoto R, Terauchi T, Nakazato Y, Kubomura K, Wada M. Determining the extent of tumor resection at surgical planning with 18F-fluciclovine PET/CT in patients with suspected glioma: multicenter phase III trials. Ann Nucl Med. 2021 Dec;35(12):1279-1292. doi: 10.1007/s12149-021-01670-z. Epub 2021 Aug 18. PMID 34406623
- [Background] Gondi V, Bradley K, Mehta M, Howard A, Khuntia D, Ritter M, Tome W. Impact of hybrid fluorodeoxyglucose positron-emission tomography/computed tomography on radiotherapy planning in esophageal and non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2007 Jan 1;67(1):187-95. doi: 10.1016/j.ijrobp.2006.09.033. PMID 17189070
- See also: Miami Cancer Institute — http://cancer.baptisthealth.net/